CLINICAL TRIAL: NCT01293474
Title: Choroidal Thickness in Glaucoma Patients and Healthy Controls
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EDI-OCT
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Glaucoma Patients and Healthy Controls
MeSH Terms: interventions — Proton Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- glaucoma patients: patients with diagnosis of primary open angle glaucoma
  Interventions: Device: Spectralis® SD-OCT, Heidelberg Engineering GmbH, H
- control group: age matched healthy controls
  Interventions: Device: Spectralis® SD-OCT, Heidelberg Engineering GmbH, H

INTERVENTIONS:
Device: Spectralis® SD-OCT, Heidelberg Engineering GmbH, H — Measurement of the choroidal thickness with Spectralis® SD-OCT

SUMMARY:
With the new software tool (EDI, enhanced depth imaging) of the Spectralis® spectral-domain optical coherence tomography (SD-OCT) it is possible to visualize and measure the choroidal thickness. In glaucoma a vascular component is known. Therefore a difference of choroidal thickness in glaucoma patients and healthy controls is proposed.

* Trial with medical device

ELIGIBILITY:
Inclusion criteria: for both groups (glaucoma study group and control group):

men and women of at least 50 years of age

for the glaucoma study group: diagnosis of primary open angle glaucoma (POAG)

Exclusion criteria: for both groups (glaucoma study group and control group):

* less then 50 years of age
* any pathology of the central retina
* any optic nerve disorder other then glaucoma
* retinal vascular disorder

for the glaucoma study group: other glaucoma diagnosis then primary open angle glaucoma

for the control group: any diagnosis of glaucoma

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients and controls are selected out of our primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
COV | t0

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kniestedt, Ass. Prof., MD, Principal Investigator — University Hospital Zurich, Ophtalmic Clinic
Locations (1):
- University Hospital Zurich, Ophthalmic Clinic, Zurich, Canton of Zurich, Switzerland